CLINICAL TRIAL: NCT06590766
Title: Impact of Acupuncture and Manual Therapies on Patients' Quality-of-life in a Hospital-to-community Continuum of Integrative Oncology and Supportive-palliative Care
Brief Title: Impact of Acupuncture and Manual Therapies on Patients' Quality-of-life in a Hospital-to-community Continuum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Director, Integrative Oncology Program, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMC-23-0004
Record Dates: First submitted 2024-08-20; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Oncology
Keywords: Integrative oncology; Palliative care; Acupuncture
MeSH Terms: conditions — Neoplasms | interventions — Acupressure; Acupuncture Therapy; Mind-Body Therapies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Integrative oncology single-modality (Experimental): Acupressure/relaxation only
  Interventions: Other: acupressure/relaxation with acupuncture
- Integrative oncology multi-modality (Experimental): Acupressure/relaxation with acupuncture
  Interventions: Other: acupressure/relaxation with acupuncture
- Palliative nursing counseling (Active Comparator): Patients choosing to undergo a palliative nursing consultation only.
  Interventions: Other: acupressure/relaxation with acupuncture

INTERVENTIONS:
Other: acupressure/relaxation with acupuncture — The acupressure/acupuncture points will be designated according to a protocol for each of the four leading concerns (pain, fatigue, emotional, and gastrointestinal), based on evidence-based research. For example, clinical guideline-based IO protocols for pain relief will include the following analgesia-related acupressure/acupuncture points: Liver-3, Taichong; Large-Intestine 4, Hegu; Stomach-36, Zusanli; Pericard-6, Neiguan; Spleen-6, Sanyinjiao; Yin tang; as well as battlefield ear acupuncture points. In both IO intervention groups, relaxation techniques will be tailored to the patient's main concern, with the option of including breathing and guided imagery modalities as well.
  Other Names: Manual and mind-body therapies

SUMMARY:
Oncology patients often suffer during hospitalization from pain, emotional distress, gastrointestinal symptoms, weakness, and quality of life (QoL)-related concerns. A large body of research has shown that acupuncture and other integrative oncology (IO) modalities, when provided in conjunction with supportive care, can significantly address and alleviate QoL-related concerns. In the proposed study, we examine an innovative model of IO and palliative care, provided to patients with cancer during hospitalization. Oncology patients at the Carmel Medical Center, Haifa, Israel, will be referred by hospital to IO/palliative care, specifying the patient's QoL-related concerns. After signing the informed consent form, patients will be asked to choose between IO intervention (Group A and B) or palliative nursing counseling only (Group C). Patients choosing to undergo integrative treatment will be randomly allocated to one of the two study interventions: acupressure-relaxation alone (Group A); or acupressure-relaxation modalities with acupuncture (Group B). The response to the study intervention for QoL-related concerns will be re-assessed immediately; at 24-48 hours; and after 2 weeks following the treatment. Patients will also undergo objective measurements during treatment using Heart Rate Variability (HRV) and Nociception Levels (NOL) to determine the impact of the intervention on their QoL and concerns. In summary, the proposed study will examine the short-term impact of an integrative/palliative intervention on patient QoL-related concerns, comparing acupressure-relaxation modalities with or without acupuncture, as well as to patients receiving palliative nursing counseling. Following discharge, treatments will be provided at one of six participating community IO services, over a 12-week period, in coordination with the oncology and palliative care teams in the community.

DETAILED DESCRIPTION:
Scientific background: The provision of complementary and integrative medicine therapies within supportive and palliative oncology care (herewith, Integrative Oncology, IO) is increasingly taking place in leading oncology centers across the globe. The Society for Integrative Oncology (SIO) and the American Society of Clinical Oncology (ASCO) have co-published clinical practice guidelines on the effective and safe use of these modalities for patients with cancer. The proposed study will explore the provision of IO care to patients with cancer during hospitalization, with the goal of addressing emotional distress, pain, fatigue, gastro-intestinal symptoms, and other quality of life (QoL)-related concerns.

Study objectives and purpose: The primary study objective is to improve patients' QoL-related concerns while hospitalized for a variety of cancer-related indications. This, in a clinical context in which in-patient IO interventions are provided together with palliative care, with the two teams coordinating their work. Secondary objective is to identify barriers and enablers to the continuity of IO care, following hospitalization, for patients with cancer, from the in-patient hospital to the out-patient community care setting.

Methods: Study design and setting: The proposed study will take place within a prospective randomized controlled methodology, beginning with a patient-preference stage, in which patients are asked to choose whether they are interested in undergoing IO treatments or palliative nursing counseling.

Study population: Patients of either gender, diagnosed with cancer, age ≥ 18 years and hospitalized in one of the five surgical/internal departments will be eligible for study inclusion. Participating patients will be referred to the study team by a medical healthcare provider in their respective departments, providing a list of clinical indications for the referral.

Allocation to study arms and groups:

Participants will be allocated to one of the two primary study arms, based on their preference for undergoing IO treatments:

* Integrative oncology (IO) arm (Groups A and B): Patients choosing to undergo IO treatments, in addition to standard palliative care
* Palliative nursing counseling (Group C): Patients choosing to undergo a palliative nursing consultation only.

Patients choosing to receive IO care will then be randomly and openly assigned to one of the intervention groups, using the "Research Randomizer" online tool (https://www.randomizer.org/), to one of the following study groups:

* Single-modality IO, receiving acupressure/relaxation only (Group A)
* Multi-modality IO receiving acupressure/relaxation with acupuncture (Group B) IO treatments and palliative nursing consultation: Patients in the intervention arm of the study (groups A and B) will be interviewed and assessed by the IO practitioner, while a palliative nurse specialist will interview those choosing the palliative nursing consultation (Group C). In all study groups, the interviews will address QoL-related concerns, identifying the patient's leading concern (e.g., pain, anxiety). Following the QOL assessment in both groups, an integrative or palliative intervention with the goal of alleviating the patient's leading QoL-related concerns over the next 24-hour period.

Patients in the IO intervention arm of the study will undergo acupressure/relaxation treatments only (Single Modality, Group A), or with the addition of acupuncture (Multi-Modality, Group B). The acupressure/acupuncture points will be designated according to a protocol for each of the four leading concerns (pain, fatigue, emotional, and gastrointestinal), based on evidence-based research. The palliative nursing intervention (Group C) will entail a personalized bio-psycho-social-oriented discussion, highlighting the patient's and their informal caregiver's unmet needs and QoL-related concerns.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with cancer, age ≥ 18 years and hospitalized in one of the six internal medicine and surgical departments in the hospital.

Exclusion Criteria:

Inability to read and provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessing patients' QoL-related concerns will be performed using the Edmonton Symptom Assessment Scale (ESAS) | Before and immediately following the IO intervention; at 24-48 hours; and two weeks post-treatment.
  Assessing the effectiveness and safety of an IO intervention involving acupressure and relaxation, either with or without the addition of acupuncture, on the severity of QoL-related concerns among hospitalized oncology patients. Of the three PROMs, ESAS asks respondents to score a list of 10 QoL-related concerns on a scale from 0 (no symptom) to 10 (worst severity of the symptom).
Assessing patients' QoL-related concerns will be performed using the Measure Yourself Concerns and Wellbeing (MYCAW). | Before and immediately following the IO intervention; at 24-48 hours; and two weeks post-treatment.
  Of the three PROMs used to assess patients' QoL, in MYCAW, patients to list and then score (from 0 to 6; 6 is most severe) their 2 most severe QoL-related concerns.
Assessing patients' QoL-related concerns will be performed using the European Organization for Research and Treatment of Cancer Quality of Life(EORTC QLQ-C30). | Before and immediately following the IO intervention; at 24-48 hours; and two weeks post-treatment.
  EORTC QLQ C-30 asks a number of QoL-related clusters of concerns, from 1 (not at all) to 4 (very much).
Assessment of objective physiological changes during the intervention | During the 30 minutes intervention
  Assessment of objective physiological changes during the 30-minute intervention will be conducted using chest-lead electrocardiogram monitoring autonomic heart rate variability (HRV) throughout. At the same time, nociceptive levels (NOL) will be monitored using a PMD-200 device (Medasense, Ramat Gan, Israel).

SECONDARY OUTCOMES:
Identifying the most commonly reported QoL-related concerns of hospitalized oncology patients. This based on the Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire. | Before and immediately following the 30-minute intervention.
  Identify and evaluating the most commonly reported QoL-related concerns of patients during hospitalization and the indications for which the hospital staff refer them to the IO treatment program. In MYCAW, patients to list and then score (from 0 to 6; 6 is most severe) their 2 most severe QoL-related concerns. In addition to quantitative assessment of patient concerns, a qualitative assessment will be performed using the MYCAW narratives as reported by patients following open-ended questions.
Identifying barriers and enablers to the continuity of integrative oncology care.This based on the Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire. | Two weeks for patients with localized cancer; 12 weeks for patients with advanced cancer
  Identifying barriers and enablers to the continuity of integrative oncology care for patients with cancer, from the in-patient hospital to the out-patient community care setting. MYCAW questionnaire include also a qualitative segment where patients are asked to report on their feedback and experience following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical center, Haifa, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao JJ, Ismaila N, Bao T, Barton D, Ben-Arye E, Garland EL, Greenlee H, Leblanc T, Lee RT, Lopez AM, Loprinzi C, Lyman GH, MacLeod J, Master VA, Ramchandran K, Wagner LI, Walker EM, Bruner DW, Witt CM, Bruera E. Integrative Medicine for Pain Management in Oncology: Society for Integrative Oncology-ASCO Guideline. J Clin Oncol. 2022 Dec 1;40(34):3998-4024. doi: 10.1200/JCO.22.01357. Epub 2022 Sep 19. PMID 36122322
- [Background] Carlson LE, Ismaila N, Addington EL, Asher GN, Atreya C, Balneaves LG, Bradt J, Fuller-Shavel N, Goodman J, Hoffman CJ, Huston A, Mehta A, Paller CJ, Richardson K, Seely D, Siwik CJ, Temel JS, Rowland JH. Integrative Oncology Care of Symptoms of Anxiety and Depression in Adults With Cancer: Society for Integrative Oncology-ASCO Guideline. J Clin Oncol. 2023 Oct 1;41(28):4562-4591. doi: 10.1200/JCO.23.00857. Epub 2023 Aug 15. PMID 37582238
- [Background] Bower JE, Lacchetti C, Alici Y, Barton DL, Bruner D, Canin BE, Escalante CP, Ganz PA, Garland SN, Gupta S, Jim H, Ligibel JA, Loh KP, Peppone L, Tripathy D, Yennu S, Zick S, Mustian K. Management of Fatigue in Adult Survivors of Cancer: ASCO-Society for Integrative Oncology Guideline Update. J Clin Oncol. 2024 Jul 10;42(20):2456-2487. doi: 10.1200/JCO.24.00541. Epub 2024 May 16. PMID 38754041